CLINICAL TRIAL: NCT00903864
Title: Blood Pressure Monitor Clinical Test (Cuff Range: 22 cm-30 cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Other Study IDs: AndonHealth1
Record Dates: First submitted 2009-05-14; First posted 2009-05-19 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Blood Pressure

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- stethoscopy
- BPM: blood pressure monitor

SUMMARY:
The purpose of this study is to monitor the blood pressure level of the patient using a cuff ranged 22 cm-30 cm.

ELIGIBILITY:
Inclusion Criteria:

* arm range: 22 cm-30 cm

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People whose arm range is 22 cm-30 cm
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual)